CLINICAL TRIAL: NCT04363099
Title: Multicentre Observational Study on Management COVID 19 Positive Outpatients in a French Cluster.
Acronym: COVID AMBU 60
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maison de Sante Pluridisciplinaire de Creil (Other)
Responsible Party: Principal Investigator, DIMI Svetlane, Dr, Maison de Sante Pluridisciplinaire de Creil
Other Study IDs: 2020-A01059-30
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: ambulatory; outpatients; COVID 19; Oise, France
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- outpatients COVID 19 positive
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — observational management of outpatients COVID 19

SUMMARY:
Since December 2019, a new agent, the coronavirus SARS-Cov-2, has spread from China to the rest of the world causing an international epidemic of respiratory diseases called COVID-19. Oise was one of the first clusters in France, with more than 4,000 confirmed cases. A significant proportion (80%) of patients with COVID-19 are ambulatory. However, few data are available for this particular population in France. Thus, few clear recommendations are available.

We propose to conduct a large cohort of observation of suspected or confirmed COVID-19 patients on an ambulatory basis in the Oise region. This observatory will make it possible to describe the epidemiological characteristics and initial management of COVID-19 patients and to identify early severity factors.

ELIGIBILITY:
Inclusion Criteria:

* patients with covid 19 symptoms
* patients who had a contact with a person PCR Covid 19+

Exclusion Criteria:

* none

Max Age: 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: ambulatory patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical description of covid 19 ambulatory cases. | 3 months

SECONDARY OUTCOMES:
Biological and radiological description of ambulatory cases | 3 months
Prevalence of positive cases (PCR and/or serological positive) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Msp de Creil, Creil, France

IPD SHARING:
Plan to Share IPD: Undecided